CLINICAL TRIAL: NCT02194270
Title: Relative Bioavailability of Ambroxol Hydrochloride Following Oral Administration of Soft Pastilles 15 mg (Test) Compared to 15 mg of Syrup (15mg/5mL, Reference I) and Compared to 15 mg of Syrup (30mg/5mL) (Reference II) in Healthy Male and Female Volunteers. An Open-label, Randomised, Single-dose, 3-way Crossover Study
Brief Title: Relative Bioavailability of Ambroxol Hydrochloride of Soft Pastilles Compared to Ambroxol Hydrochloride Syrup in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18.488
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- Ambroxol hydrochloride - soft pastille (Experimental)
  Interventions: Drug: Ambroxol hydrochloride - soft pastille
- Ambroxol hydrochloride - syrup - low dose (Active Comparator)
  Interventions: Drug: Ambroxol hydrochloride - syrup - low dose
- Ambroxol hydrochloride - syrup - high dose (Active Comparator)
  Interventions: Drug: Ambroxol hydrochloride - syrup - high dose

INTERVENTIONS:
Drug: Ambroxol hydrochloride - soft pastille
  Arms: Ambroxol hydrochloride - soft pastille
Drug: Ambroxol hydrochloride - syrup - low dose
  Arms: Ambroxol hydrochloride - syrup - low dose
Drug: Ambroxol hydrochloride - syrup - high dose
  Arms: Ambroxol hydrochloride - syrup - high dose

SUMMARY:
Study to investigate the relative bioavailability of ambroxol hydrochloride soft pastilles 15 mg vs. ambroxol hydrochloride (HCL) 15 mg of syrup (15mg/5mL, Reference I) and ambroxol hydrochloride 15 mg of syrup (30mg/5mL, Reference II) in a fasted state

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests
* No finding deviating from normal and of clinical relevance
* No evidence of a clinically relevant concomitant disease
* Age ≥18 and Age ≤55 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. oral contraceptives, sterilization, intrauterine device (IUD)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2004-09; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 30 hours after each drug administration
Cmax (maximum concentration of the analyte in plasma) | up to 30 hours after each drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 30 hours after each drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 30 hours after each drug administration
λz (terminal rate constant in plasma) | up to 30 hours after each drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 30 hours after each drug administration
MRTpo (mean residence time of the analyte in the body after p.o. (oral) administration) | up to 30 hours after each drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 30 hours after each drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 30 hours after each drug administration
Number of patients with adverse events | up to 40 days
Number of patients with abnormal changes in laboratory parameters | up to 40 days
Number of patients with clinically significant changes in vital signs (BP (Blood pressure), PR (Pulse rate)) | up to 40 days
Assessment of tolerability by investigator on a 4-point scale | within 8 days after last administration